CLINICAL TRIAL: NCT06996210
Title: Efficacy of Acupuncture in Treating Comorbid Chronic Nonspecific Neck Pain and Insomnia
Brief Title: Effect of Acupuncture on Chronic Nonspecific Neck Pain and Insomnia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Liu Zhishun, professer, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-090-KY
Record Dates: First submitted 2025-05-14; First posted 2025-05-30 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Neck Pain Chronic; Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture group (Experimental): Participants in the acupuncture group will receive treatment at DU 20 [Baihui], EX-HN15 [Jingbailao], GB 12 [Wangu], Shangyintang (On the head, 1 B-cun superior to Yintang), HT7 [Shenmen], KI 3 [Taixi] and Ashi Point.
  The treatment will last 30 minutes for each session, 3 sessions per week (ideally every other day) for a succession of 4 weeks.
  Interventions: Device: Acupuncture
- Sham acupuncture (SA) group (Sham Comparator): Participants in the SA group will receive treatment at sham DU 20, sham EX-sham HN15, sham GB 12, sham Shangyintang , sham HT7 and sham KI 3. The treatment will last 30 minutes for each session, 3 sessions per week (ideally every other day) for a succession of 4 weeks.
  Interventions: Device: sham acupuncture

INTERVENTIONS:
Device: Acupuncture — The needles will be inserted to 12.5-30 mm in acupoints through adhesive pads. Needles will be lifted, thrusted and twirled gently for 3 times to achieve deqi sensation and manipulated every ten minutes.
  Arms: acupuncture group
Device: sham acupuncture — The needle will be inserted to 2-3mm in sham Baihui acupoint. For the remaining sham acupoints, needles will be inserted into the pad and reaching the skin. Needles will be lifted, thrusted and twirled gently for 3 times to simulate the effect of the needle tip penetrating the skin.
  Arms: Sham acupuncture (SA) group

SUMMARY:
The study aims to assess the efficacy and safety of acupuncture among patients with chronic nonspecific neck pain and insomnia, compared with sham acupuncture.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years old;
2. Meet the diagnostic criteria for both chronic nonspecific neck pain and chronic insomnia;
3. The patient's average 24-hour overall neck pain intensity score on the NRS is ≥3;
4. The patient's Insomnia Severity Index (ISI) score is ≥10;
5. The patient is willing to participate in the study and has signed the informed consent form.

Exclusion Criteria:

1. Specific neck pain with a clear etiology, including trauma, tumor, connective tissue disease, rheumatic disease, metabolic and endocrine disorders, neuropathy, spinal cord disease, fracture, or vertebral misalignment;
2. Positive Spurling test, neck flexion test, upper limb traction test, or foraminal distraction test. Neck pain accompanied by radiating pain in the upper limbs or radicular compression symptoms, or acute exacerbation of neck pain;
3. Neck pain accompanied by sensory disturbances or other neurological symptoms, or ankylosis of the facet joints;
4. Previous history of cervical spine surgery;
5. Previous history of head and neck trauma, such as whiplash injury;
6. Insomnia caused by medications (e.g., caffeine, corticosteroids), withdrawal reactions, or other underlying conditions (e.g., hyperthyroidism, severe anxiety/depressive disorders);
7. Long-term use of analgesics, muscle relaxants, or hormones, or presence of other pain more severe than neck pain;
8. Other sleep disorders, such as sleep apnea syndrome, or shift workers;
9. Presence of psychiatric disorders (e.g., depression), cognitive impairment, or language disorders;
10. Patients with drug dependency;
11. Received acupuncture treatment within the past month;
12. Severe cardiovascular, hepatic, renal, hematologic, autoimmune diseases, infectious diseases, poor general nutritional status, malignancy, or patients in the terminal stage of severe illness;
13. Pregnant or planning to become pregnant within the next year, breastfeeding, or postpartum ≤12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-27 (Estimated); Study Completion 2028-03-27 (Estimated)

PRIMARY OUTCOMES:
The change in average 24h overall neck pain intensity measured by NRS from baseline over the past week | week 5
  The NRS score ranges from 0 to 10, with higher scores indicating more severe pain.
The change from baseline in the Chinese version of the Insomnia Severity Index (ISI-C) scores. | week 5
  The Chinese version of the Insomnia Severity Index (ISI-C) will be used to assess the severity of patients' self-perceived insomnia symptoms. Each item is rated on a scale from 0 to 4, with a total score ranging from 0 to 28. Based on the total score, the severity of insomnia can be categorized into four levels: a score of 0-7 indicates "no clinically significant insomnia," 8-14 indicates "subclinical insomnia," 15-21 indicates "clinical insomnia (moderate)," and 22-28 indicates "clinical insomnia (severe)."

SECONDARY OUTCOMES:
The change in average 24h overall neck pain intensity measured by NRS from baseline over the past week | week 9 and 16
  The NRS score ranges from 0 to 10, with higher scores indicating more severe pain.
The change from baseline in the ISI-C scores. | week 9 and 16
  The ISI-C will be used to assess the severity of patients' self-perceived insomnia symptoms. Each item is rated on a scale from 0 to 4, with a total score ranging from 0 to 28. Based on the total score, the severity of insomnia can be categorized into four levels: a score of 0-7 indicates "no clinically significant insomnia," 8-14 indicates "subclinical insomnia," 15-21 indicates "clinical insomnia (moderate)," and 22-28 indicates "clinical insomnia (severe)."
The proportion of participants with at least 30% reduction in NRS scores from baseline | week 5, 9 and 16
  The NRS score ranges from 0 to 10, with higher scores indicating more severe pain.
The proportion of participants with at least 6 points reduction in ISI-C scores from baseline | week 5, 9 and 16
  The ISI-C will be used to assess the severity of patients' self-perceived insomnia symptoms. Each item is rated on a scale from 0 to 4, with a total score ranging from 0 to 28. Based on the total score, the severity of insomnia can be categorized into four levels: a score of 0-7 indicates "no clinically significant insomnia," 8-14 indicates "subclinical insomnia," 15-21 indicates "clinical insomnia (moderate)," and 22-28 indicates "clinical insomnia (severe)."
The change from baseline in the total score of the Neck Disability Index (NDI). | week 5, 9 and 16
  Neck Disability Index (NDI) consists of 10 items, with a total score ranging from 0 to 50. A higher score indicates a greater impact of neck pain on quality of life.
The proportion of participants with at least 10 points reduction in NDI scores from baseline | week 5, 9 and 16
  NDI consists of 10 items, with a total score ranging from 0 to 50. A higher score indicates a greater impact of neck pain on quality of life.
The change from baseline in the maximum pain intensity score on the NRS during six directions of neck movement. | week 5, 9 and 16
  The NRS score ranges from 0 to 10, with higher scores indicating more severe pain.
The change from baseline in the Pittsburgh Sleep Quality Index (PSQI). | week 5, 9 and 16
  The PSQI has a total score ranging from 0 to 21. A higher score indicates poorer sleep quality. Specifically, a total score of 0-5 indicates very good sleep quality; 6-10 indicates fairly good sleep quality; 11-15 indicates average sleep quality; and 16-21 indicates poor sleep quality.
The change from baseline in the Hospital Anxiety and Depression Scale (HADS) scores. | week 5, 9 and 16
  The HADS score ranges from 0 to 42, with higher scores indicating greater anxiety and depression.
The proportion of responders per the Patient Global Impression of Change (PGI-C) | week 5 and 16
  The PGI-C evaluates the overall treatment effect perceived by patients themselves. The change can be rated in 7 levels, including "very much better", "moderately better, "a little better", "no change", "a little worse", "moderately worse" or "very much worse".
The percentage of patients who used rescue analgesics and sedative-hypnotics. | week 5, 9 and 16
  The percentage of patients who used emergency analgesics and sedative-hypnotics.
The total number of days of using rescue analgesics and sedative-hypnotics. | week 5, 9 and 16
  The total number of days of using rescue analgesics and sedative-hypnotics.
Blinding assessment | Within 5 minutes after the last treatment at week 4.
  In this trial, two types of acupuncture treatments were used: traditional acupuncture, which has a stronger sensation of needle insertion, and modern acupuncture, which has a weaker sensation of needle insertion. Patients were asked which type of therapy they thought they had received.

OTHER OUTCOMES:
Expectance assessment | baseline
  Patients wIll be asked to predict how their chronic neck pain will change in one month (much better, somewhat better, uncertain, somewhat worse, much worse); and how their insomnia will change (much better, somewhat better, uncertain, somewhat worse, much worse).
Incidence of advers events | through study completion, an average of 16 weeks
  Adverse events and severe adverse events will be recorded in the case report form, whether related to interventions or not.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences; Guangxia Shi, Principal Investigator — Beijing University of Chinese Meidicine

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data and data dictionary will be available with the publication until six months after publication.
  A formal request should be sent to zhishunjournal@163.com with a methodologically sound proposal.
  Researchers whose proposal has been approved will sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available with the publication until six months after publication.
Access Criteria: A formal request should be sent to zhishunjournal@163.com with a methodologically sound proposal. Researchers whose proposal has been approved.
  Researchers whose proposal has been approved will sign a data access agreement.